CLINICAL TRIAL: NCT03434912
Title: Identification and Evaluation of the Potential Biomarkers on Circulating Tumor Cells and Tumor Related Rare Cells in Cancer Patients Undergoing Immunotherapy
Brief Title: Identification and Evaluation of Circulating Tumor Cells and Tumor Related Rare Cells in Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MiCareo Taiwan Co., Ltd. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: MiC-SRS-HNSCC-001
Record Dates: First submitted 2018-02-07; First posted 2018-02-15 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-05

CONDITIONS: CTC and Tumor Related Rare Cell
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is designed to evaluate the enumeration of circulating tumor cells and identify the potential biomarkers associated with clinical outcome. The secondary objective is to explore whether the changes of tumor related rare cells associates clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Over 20 years of age.
3. Cancer patients on immune checkpoint inhibitors.

Exclusion Criteria:

1. Subjects who have other cancer history
2. Pregnant females
3. Subjects with active, known or suspected autoimmune disease.
4. Known history of human immunodeficiency virus (HIV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 cancer patients undergoing immunotherapy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cell | 1 years
  Isolation and analysis of circulating tumor cells before and after immunotherapy

SECONDARY OUTCOMES:
tumor related rare cell | 1 years
  Isolation and analysis of tumor related rare cells before and after immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan